CLINICAL TRIAL: NCT05152394
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Exosome Intranasal Instillation for the Treatment of Parkinson's Disease
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Exosomes for Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-016
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; stem cell treatment
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloEx) (Experimental): Intranasal instillations of 4 CCs of AlloEx, approximately 800 billion exosomes. Treatments on back-to-back days, totaling 2 doses.
  Interventions: Biological: AlloEx

INTERVENTIONS:
Biological: AlloEx — cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes

SUMMARY:
This trial will study the safety and efficacy of intranasal instillation of cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes for the treatment of Parkinson's Disease

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of intranasal installation of cultured allogeneic adult umbilical cord derived mesenchymal stem cell (UC-MSC) exosomes for the treatment of Parkinson's Disease. Patients will receive a dose of 4 CCs of AlloEx, approximately 800 billion exosomes, between both nasal cavities. A second equivalent dose will be administered on the subsequent day. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur
* Anticoagulation medicine use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No